CLINICAL TRIAL: NCT00175409
Title: Breast Feeding Analgesia in Preterm Infants
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: University of British Columbia (Other)
Collaborators: SickKids Foundation (Other)
Responsible Party: Dr. Liisa Holsti, University of British Columbia
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: C05-0248
Record Dates: First submitted 2005-09-11; First posted 2005-09-15 (Estimated); Last update posted 2011-04-12 (Estimated); Status verified 2011-04

CONDITIONS: Pain
Keywords: Pain Response
MeSH Terms: conditions — Pain | interventions — Blood Specimen Collection

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- 1 (Active Comparator): Infants will be randomized to two interventions which will take place during two separate blood collections that are required for clinical management. For the standard care condition, infants will remain in their isolettes and will be positioned in prone and given a pacifier to suck on throughout the blood collection.
  Interventions: Procedure: Blood collection
- 2 (Active Comparator): Infants will be randomized to two interventions which will take place during two separate blood collections that are required for clinical management. For the feeding condition, infants will be held and then breast fed by their mother during the blood collection.
  Interventions: Procedure: Blood collection

INTERVENTIONS:
Procedure: Blood collection — For the standard care condition, infants will remain in their isolettes and will be positioned in prone and given a pacifier to suck on throughout the blood collection.
  Arms: 1
Procedure: Blood collection — For the feeding condition, infants will be held and then breast fed by their mother during the blood collection.
  Arms: 2

SUMMARY:
The purpose of this study is to compare the effects of mothers' breastfeeding with the effects of pacifier sucking on preterm infant biobehavioural responses during and immediately after a painful procedure

Hypothesis:

1. When breast fed by their mothers during blood collection, preterm infants will show less pain reaction than when sucking on a pacifier.
2. Following breast feeding during the blood collection, mothers will find no differences in their infants' breast feeding ability.

DETAILED DESCRIPTION:
Research Method:

In a within subjects, randomized, cross-over design, 50 stable preterm infants born between 30-36 weeks gestational age will be studied. Infants will be randomized to two interventions which will take place during two separate blood collections that are required for clinical management. For the standard care condition, infants will remain in their isolettes and will be positioned in prone and given a pacifier to suck on throughout the blood collection. For the feeding condition, infants will be held and then breast fed by their mother during the blood collection.

ELIGIBILITY:
Inclusion Criteria:

* born between 30-36 weeks gestational age
* breastfeeding
* mother has fluent English

Exclusion Criteria:

* CNS injury
* congenital anomaly
* active infection
* has had surgeries or analgesics/sedatives in last 72 hours
* history of maternal drug exposure

Ages: 3 Days to 37 Weeks | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 50 (Estimated)
Dates: Start 2008-01; Primary Completion 2010-06 (Actual); Study Completion 2010-06 (Actual)

PRIMARY OUTCOMES:
Videotaped and recorded at Baseline, Lance and Recovery:
Behavioral Indicators of Infant Pain (BIIP) - total score
Heart Rate

SECONDARY OUTCOMES:
Videotaped and Recorded at Baseline, Lance and Recovery:
Hand Movements
Sleep/Wake States
Samples taken at baseline, lance and recovery
Salivary Cortisol sample
Recorded before the breast feeding intervention and at 24 hours following:
Preterm Infant Breastfeeding Behavior Scale

CONTACTS AND LOCATIONS:
Overall Officials: Liisa Holsti, PhD, OT, Principal Investigator — University of British Columbia
Locations (2):
- Canada (2):
  - Lions Gate Hospital - Special Care Nursery, North Vancouver, British Columbia
  - Children's and Women's Health Centre of British Columbia - Neonatal Intensive Care Unit & Intermediate Care Nursery, Vancouver, British Columbia